CLINICAL TRIAL: NCT07340957
Title: Validation of the B. Well Digital Upper Arm Blood Pressure Monitor Pro-25 According to ISO 81060- 2
Brief Title: Valid-B.Well BP25 Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: B.Well Swiss AG (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BWE-01
Record Dates: First submitted 2025-11-26; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Volunteers; Study Focus: Blood Pressure Measures
Keywords: blood pressure; iso 81060-2; upper arm blood pressure monitor; commercialized device validation
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-arm, open, comparative, validation of a commercialized device, with repeated measures accuracy study designed in accordance with the requirements of the ISO 81060-2:2018 AAMI/ESH/ISO Universal Standard for the clinical validation of automated non-invasive sphygmomanometers (Non-invasive sphygmomano-meters - Part 2: Clinical investigation of intermittent automated measurement, including Amendments 1 and 2)).
  The study aims to clinically evaluate the accuracy of the B-Well PRO-25 upper arm automated sphygmomanometer for systolic blood pressure (SBP) and diastolic blood pressure (DBP) in adults and adolescents in accordance with ISO 81060-2.
  The comparative measurements are obtained through auscultation by an observer using a mercury sphygmomanometer (reference method).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sigle arm (Experimental): Single-arm. All subjects will undergo blood pressure measurement with the reference manual method and with upper arm automated sphygmomanometer (3 times each).
  Interventions: Diagnostic Test: Blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Blood pressure measurement — All measurements will be performed by trained observers in line with the requirements of the ISO 81060-2:2018 AAMI/ESH/ISO Universal Standard (1), ensuring accuracy, consistency, and reproducibility.
  The investigation shall be performed in an isolated room under comfortable ambient temperature.
  * The cuff shall be applied on the bare arm with no compression proximal to the cuff.
  * The subject shall rest quietly for at least 10 minutes prior to the start of measurements.
  * The subject should avoid talking during the entire measurement procedure.
  * BP shall be measured on the subject's left arm at heart level.
  * A minimum of 5 minutes shall elapse prior to obtaining the first reference blood pressure measurement.

SUMMARY:
Prospective, single-center, single-arm, open, comparative, validation of a commercialized device, repeated measures accuracy study designed in accordance with the requirements of the ISO 81060-2:2018 AAMI/ESH/ISO Universal Standard for the clinical validation of automated non-invasive sphygmomanometers (Non-invasive sphygmomano-meters - Part 2: Clinical investigation of intermittent automated measurement, including Amendments 1 and 2)).

The validation will be conducted with volunteers rather than necessarily with patients, and all measurements will be performed outside of the subjects' normal diagnosis or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 years
* Signed Informed Consent

Exclusion Criteria:

* Any medical condition preventing light to moderate arm compression
* Absence of the upper arm
* Subjects with upper arm circumference <22 cm or >42 cm
* Subjects with severe shock;
* Subjects with a history of mental illness or current mental disorders;
* Patients with arrhythmias (atrial premature beats, ventricular premature beats, atrial fibrillation, etc.) or upper limb arteriosclerosis (at the direct measurement site);
* Subjects using extracorporeal circulation devices;
* Subjects with excessive limb asymmetry;
* Subjects who have undergone mastectomy or lymph node dissection;
* Subjects with arm injuries or exposed wounds, or those with circulatory disorders;
* Subjects with vascular accesses in the arms or arteriovenous shunt tubes;
* Subjects who have participated in other clinical trials within the past 1 month;
* Subjects for whom the procedures during the clinical trial may pose excessive medical risks;
* Subjects determined by the investigator to be unsuitable for participating in the clinical study.
* Subject under judicial protection, guardianship or curatorship or participant deprived of their liberty by judicial or administrative decision

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The study will assess compliance with the following validation criteria defined by the standard ISO 81060-2:2018: Criterion 1 - Group-level accuracy (paired-difference analysis). Criterion 2 - Subject-level accuracy | Day 1
  The study will assess compliance with the following validation criteria defined by the standard ISO 81060-2:2018 for SBP and DBP (in mmHg):
  Criterion 1 - Group-level accuracy (paired-difference analysis). For systolic blood pressure (SBP) and diastolic blood pressure (DBP) separately, the mean difference between the test device and the reference method (observer auscultation with a mercury sphygmomanometer) across all valid paired determinations shall be within ±5 mmHg, and the standard deviation (SD) of these differences shall be ≤ 8 mmHg.
  Criterion 2 - Subject-level accuracy For SBP and DBP, each subject's mean difference (test device - reference) shall be calculated from that subject's repeated paired determinations. The standard deviation of these subject-level means across all subjects shall comply with the requirements specified in Table 1 Averaged subject data acceptance in mmHg of ISO 81060-2:2018 (1) for SBP and DBP.

SECONDARY OUTCOMES:
Agreement by Bland-Altman analysis | Day 1
  Calculation of the bias (average difference between test device and reference method) and the 95% limits of agreement (LoA) for systolic blood pressure (SBP) and diastolic blood pressure (DBP), overall and across the blood pressure range
Population characteristics- Age | Day 1
  Age (descriptive summary)
Population Characteristics - Sex | day 1
  Sex (descriptive summaries)
Population Characteristics- arm circumferences | Day 1
  arm circumferences (descriptive summaries)
Population Characteristics- baseline blood pressure categories | Day 1
  Normotensive/hypertensive ranges for both systolic and diastolic pressures
Observser agreement | Day 1
  percentage of paired measurements (within +/- 4 mmHg)

IPD SHARING:
Plan to Share IPD: Undecided